CLINICAL TRIAL: NCT04115657
Title: The Effect of Different Starches of Boba Pearls and Sugar Substitutes Used in Milk Tea on Glycaemia, Insulinaemia and Appetite Control (Pearl Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2018/01194
Record Dates: First submitted 2019-10-03; First posted 2019-10-04 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Diabete Type 2; Obese
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — starch synthase IV, Arabidopsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Starch 1 (Experimental): Tapioca starch
  Interventions: Other: Starch 1
- Starch 2 (Experimental): High amylose
  Interventions: Other: Starch 2
- Starch 3 (Experimental): Kithul flour
  Interventions: Other: Starch 3
- Starch 4 (Experimental): Sago flour
  Interventions: Other: Starch 4
- Sugar 1 (Experimental): Pure palatinose
  Interventions: Other: Sugar 1
- Sugar 2 (Experimental): Blend of sucrose and palatinose
  Interventions: Other: Sugar 2

INTERVENTIONS:
Other: Starch 1 — Consumption of milk tea with sucrose and boba pearls made from tapioca starch
  Arms: Starch 1
Other: Starch 2 — Consumption of milk tea with sucrose and boba pearls made from high amylose
  Arms: Starch 2
Other: Starch 3 — Consumption of milk tea with sucrose and boba pearls made from kithul flour
  Arms: Starch 3
Other: Starch 4 — Consumption of milk tea with sucrose and boba pearls made from sago flour
  Arms: Starch 4
Other: Sugar 1 — Consumption of milk tea with pure palatinose and boba pearls made from tapioca starch
  Arms: Sugar 1
Other: Sugar 2 — Consumption of milk tea with blend of sucrose and palatinose and boba pearls made from tapioca starch
  Arms: Sugar 2

SUMMARY:
The first objective is to investigate the effect of boba pearls made from different starches on glycaemia, insulinaemia and appetite control. The second objective is to investigate the effects of various sugar blends of sucrose with sugar substitutes in milk tea on glycaemia, insulinaemia and appetite control.

DETAILED DESCRIPTION:
Design: There are two parts to this study. Participants will voluntarily choose to participate in either one or both parts of the study during the first screening session. Part A: Testing the effects of boba pearls using different starches. Part B: Testing the effects of milk-based tea with different sugar blends of sucrose with sugar substitutes with a standard type of boba pearl

Both parts of the study will have a randomized, nonblinded, crossover design. Screening will occur before the study commences. Participants will be asked to return on four non-consecutive days (Part A) and two-three non-consecutive days (Part B) with a wash out period of at least 2 days to avoid crossover effects. In both parts of the study, the test foods will be consumed with a carbohydrate-based food (for example: bread, biscuit etc.)

Study protocol Screening session: All potential participants will be asked to attend one screening session to ensure they are eligible to be enrolled into the study. After which, they will attend either four test sessions (Part A) and/or two-three test sessions (Part B). If the participant participates in Part A of the study, they will only be required to attend two test sessions in Part B as they would have completed the control session in Part A. If participants decide to participate only in Part B of the study, they will have to complete three test sessions. During the first screening session, participants will receive an informed consent form and be given ample time to go through it and rectify any queries they have. If they decide to take part in the study, they will be asked to sign the informed consent form. They will then be asked to complete a screening questionnaire, baseline measurements including anthropometric measurements, blood pressure, and fasting blood glucose will be collected from each participant in order to determine their eligibility. During the test sessions, participants' glycaemic, insulinaemic and appetite responses to the test meals will be measured. The test duration for each session will be 4 hours. Participants will be instructed to avoid strenuous physical activity for at least 3 days and avoid caffeine and alcohol consumption for at least 1 day prior to visiting the CNRC for their study trials. Participants will be provided with a standardised dinner meal (consisting of rice/noodles, vegetables, meat, drink/pudding) and asked to refrain from alcohol and exercise the day before their testing sessions. Screening questionnaire: The screening questionnaire will include contact information, demographic and general health details. This information will be used to determine whether the participant is eligible for the study, as well as to check for any possible confounders that may influence the study outcomes.

Anthropometric measurements: Body weight and body composition will be measured using bioelectrical impedance analysis. Height will be measured using a stadiometer in order to calculate participants' BMI. Blood pressure will also be measured. All measurements will be taken in duplicate during the screening session. Waist circumference will be measured at the minimum circumference between the iliac crest and the rib cage. Hip circumference will be measured at the maximum protuberance of the buttocks. Biceps and triceps skinfold measurements will also be taken. Blood pressure will be measured using an Omron blood pressure monitor (Model HEM-907) at baseline. Participants will be seated for five minutes before blood pressure is measured. Measurements will be taken in duplicate and the averaged results will be recorded.

Blood collection: Participants will be asked to attend the testing sessions after an overnight fast of ten hours. After a 15-minute rest period, they will have a cannula inserted in their arm to obtain blood samples at regular intervals. One fasting blood sample will be collected by venous cannulation. 3 millilitres (ml) of venous blood will be collected into Vacutainers® (Belton Dickinson Diagnostics) containing disodium EDTA for the analyses of plasma glucose, insulin concentrations. Participants will then consume treatment meal within15 minutes. Blood samples will be taken at 15, 30, 45, 60, 90, 120, 150 and 180 minutes. The amount of blood that will be collected at every time point will be about 0.6 teaspoon of blood (approximately 3 ml). The accumulative amount per test session will not be more than 5.4 teaspoons of blood (approximately 27 ml), and the accumulative amount for the entire study duration will be approximately 108ml of blood for Part A and for Part B, 81ml of blood (3 test sessions) or 54ml of blood (2 test sessions). The blood samples collected at each time point will be measured for glucose and insulin. Glycaemic and insulinaemic responses will be determined using the method described by Wolever and Jenkins. The area under the curve will be determined as the area of those increments above baseline only. Metabolic satiety: At the same time intervals, the participants will be instructed to fill in visual analogue scale (VAS) on feelings of fullness, hunger, desire to eat and prospective food consumption. VAS are 100 mm continuous lines anchored with opposing answers to a specific question asked either on a computer or on a hard copy. The specific questions asked will be, 'How hungry do you feel?', 'How full do you feel?', 'How strong is your desire to eat?', 'How much more food do you think you can eat?'. The participants will be instructed to make a mark on the line which corresponds with their subjective feeling. Only for Part A of the study, upon completion of the blood collection and before lunch, participants will be asked to drink a mouthful of the bubble tea with pearls (standardised serving size) and to masticate the boba pearls as they would naturally do. They will be asked to raise their hands once they swallow the pearls. The researcher would have counted the number of chews (x chews) to reach the swallow point (when participants raise their hands). Participants will be asked to rinse their mouth, have the second mouthful and chew x times before expectorating the bolus for particle size analysis. Three replicates will be collected. Boluses will be placed in a petri dish and suspended in distilled water to separate the particles before an image is captured for image analysis. Samples will be discarded upon completion of image analysis.

Test session: Participants will be provided a standard dinner meal to be consumed at home at 7pm the night before the test session on the day of screening for the first session. For subsequent sessions, all standard dinners will be provided on the last day of each session to be eaten before the next session. The foods are frozen dinners and can be stored in the freezer and then reheated to be consumed before the next session. After which, they will be asked to not eat and drink anything except water after 10:30 pm. They will also be instructed to arrive at the CNRC the following morning after an overnight fast of 10-12 hours. After 15 minutes upon arrival, an indwelling catheter will be inserted into a vein in your forearm and will be kept patent (free of clots) for the remainder of the test session. We will then take a blood sample from the cannula to measure baseline values. After obtaining the baseline blood samples, participants will be given the test meal to consume within 15 minutes. Following the test meal, we will take further blood samples (from the cannula) for the next 15, 30, 45, 60, 90, 120, 150 and 180 minutes. Participants will also be asked to complete the VAS following the same time points from baseline to 180 minutes. After 3 hours, the cannula will be removed and for Part A of the study, participants will be instructed to masticate boba pearls and the number of chews to reach swallow point will be recorded. Boluses of the pearls will be collected and kept for analysis. For both Part A and B, they will then be asked to consume an ad libitum lunch until they are comfortably full. At the end of the ad libitum lunch, participants will be asked to complete a final VAS for the measurement of hunger and feelings of fullness. After which, they are free to leave CNRC. During the entire testing period the participants will be instructed to remain rested and in the laboratory. There will be no incidental findings as analysed samples are basic metabolites and therefore, reporting is not applicable.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Healthy Asian Chinese
* Aged between 21 - 40 years
* ≥45kg body weight
* Body mass index between 18.5 to 25.0 kg/m2
* Normal blood pressure ≤140/90 mmHg
* Fasting blood glucose <5.6 mmol/L

Exclusion Criteria:

* Smoking
* Allergic/intolerant to any of the test foods to be administered, or any of the following common food and ingredients: eggs, fish, milk, peanuts, tree nuts, shellfish, soya, wheat, gluten, cereal, fruits, dairy products, meat, vegetable, sugar and sweetener, natural food colourings or flavourings, sulphites etc.
* Anyone with intentional food restrictions
* People with known glucose-6-phosphate dehydrogenase deficiency (G6PD deficiency)
* Having metabolic or cardiovascular diseases (such as diabetes, hypertension, heart condition, etc.)
* Having medical conditions and/or taking medications known to affect glycaemia (glucocorticoids, thyroid hormones, thiazide diuretics)
* Taking any prescribed medication or dietary supplements which may interfere with the study measurements
* Individuals who have any major organ dysfunction (eg. cardiovascular, respiratory, hepatic, renal, gastrointestinal) that may influence taste, olfaction, appetite, digestion, metabolism, absorption or elimination of test foods, nutraceutical or drug
* Excessive alcohol consumption: consuming ≥ 6 alcoholic drinks per week
* Have known Chronic infection or known to suffer from or have previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV)
* Have active Tuberculosis (TB) or currently receiving treatment for TB
* Individuals who partake in sports at the competitive and/or endurance levels
* A team member of the study or is an immediate family member (Immediate family defined as a spouse, parent, child, or sibling, whether biological or legally adopted)

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All healthy male volunteers
Enrollment: 12 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose | From 0 to 180 minutes
  Venous blood plasma measured using the COBAS
Postprandial insulin | From 0 to 180 minutes
  Venous blood plasma measured using the COBAS

SECONDARY OUTCOMES:
Appetite control | From 0 to 180 minutes
  Visual analogue scale measurement and ad libitum lunch

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No